CLINICAL TRIAL: NCT01446016
Title: Phase II Study of The Efficacy And Safety of Chloroquine (C) in CombinAtion With Taxane or Taxane-like (T) Chemo Agents in The Treatment of Patients With Advanced or Metastatic Breast Cancer Who Have Failed Anthracycline Chemo Base Therapy
Brief Title: Chloroquine With Taxane Chemotherapy for Advanced or Metastatic Breast Cancer After Anthracycline Failure (CAT)
Acronym: CAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Jenny C. Chang, MD, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00006423; 0811-0147 (Other: HMRI IRB)
Record Dates: First submitted 2011-09-29; First posted 2011-10-04 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Breast Neoplasms; Breast Cancer
Keywords: Breast Cancer; Breast Tumors; Cancer of Breast; Cancer of the Breast; Human Mammary Carcinoma; Mammary Carcinoma, Human; Mammary Neoplasm, Human; Mammary Neoplasms, Human; Neoplasms, Breast; Tumors, Breast; Chloroquine; Paclitaxel; Taxol; Ixabepilone; Abraxane; Metastatic Breast Cancer; Advanced Breast Cancer; Anthracycline
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; taxane; Docetaxel; Albumin-Bound Paclitaxel; ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chloroquine with Taxane or Taxane-Like (Paclitaxel, Docetaxel, Abraxane, Ixabepilone) Chemotherapy (Experimental): Chloroquine (250 mg) was given daily orally with either Paclitaxel or Docetaxel or Abraxane or Ixabepilone chemotherapy every 3 weeks (1 cycle) fro a maximum of 6 cycles.
  Interventions: Drug: Paclitaxel; Drug: Docetaxel; Drug: Abraxane; Drug: Ixabepilone

INTERVENTIONS:
Drug: Paclitaxel — Chloroquine 250mg po daily together with Paclitaxel (Taxane) 175 mg/m2 three hours infusion every three weeks.
  Other Names: Taxane
Drug: Docetaxel — Chloroquine 250mg po daily together with docetaxel 75 mg/m2 administered intravenously over one hour every three weeks
  Other Names: Taxane
Drug: Abraxane — Chloroquine 250mg po daily together with Abraxane 260 mg/m2 administered intravenously over 30 minutes every three weeks.
  Other Names: Taxane-like
Drug: Ixabepilone — Chloroquine 250mg po daily together with Ixabepilone is 40 mg/m2 administered intravenously over three hours every three weeks.
  Other Names: Taxane-like

SUMMARY:
The major purpose of this research study is to better understand how therapy works on different patients. This study is being offered to patients with a diagnosis of advanced or metastatic breast cancer who have failed anthracycline based therapy.

The investigators want to see the response of breast cancer cell when treated with Chloroquine used in combination with chemotherapy. Chemotherapy is an anti-cancer drug that is given through your vein. The chemotherapy used in this study is either Taxane (Paclitaxel) or Taxane-like drugs (Abraxane, Ixabepilone or Docetaxel).

DETAILED DESCRIPTION:
The purpose of this study is to determine the anti-tumor activity of the combination of Chloroquine combined with a Taxane or Taxane-like chemo agents(Paclitaxel, Docetaxel, Abraxane, Ixabepilone).

The laboratories have developed robust preclinical models utilizing both in vitro systems such as the mammosphere (MS) culture and in vivo systems such as human breast cancer xenografts allowing the investigators to identify agents which selectively target TICs, as single agents or in combination. These models are critical since tumor initiating cells (TICs) comprise only a small percentage of the tumor bulk, so that clinical tumor regression may not be observed with inhibitors that selectively target TIC self-renewal alone. Nonetheless, these agents in combination with conventional therapy may effectively kill both actively cycling or fully differentiated cells and the TIC subpopulation, leading to long term remission and eradication of cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. Females with pathologically determined advanced or metastatic breast cancer.
2. Have progressed after treatment with regimen that included an anthracycline.
3. Have had at least 4 cycles of an anthracycline containing regimen or 2 cycles if progressing on treatment.
4. Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors.
5. ≥18 years of age.
6. ECOG PS of 0, 1, or 2.
7. Laboratory values within the following ranges:

   * Hemoglobin ≥9.0gm/dL (≥1.5μmol/L); transfusions permitted.
   * Absolute neutrophil count ≥1500/mm3 (1.5 x 109/L)
   * Platelet count ≥100,000/mm3 (100 x 109/L)
   * Creatinine (Cr) <2 X the upper limit of normal (ULN), Cr clearance (CrCl) ≥30 by Cockcroft and Gault
   * Alanine aminotransferase and aspartate aminotransferase <2 X the ULN; if liver metastases are present then must be <5 X the ULN, Bilirubin <2 X the ULN, Potassium within normal limits, Magnesium within normal limits
8. Negative serum pregnancy test at the time of first dose for women of childbearing potential (WOCBP). For WOCBP, adequate contraception must be used throughout the study. For this study, acceptable methods of contraception include a reliable intrauterine device or a spermicide in combination with a barrier method. Women who are already on hormonal forms of birth control may continue that treatment but must also use a barrier method.
9. Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments.
10. Patient must be willing to undergo breast biopsies as required by the study protocol.

Exclusion Criteria:

1. Radiation therapy within 2 weeks; or chemotherapy or non-cytotoxic investigational agents within 4 weeks of initiating study treatment.
2. Evidence of New York Heart Association class III or greater cardiac disease.
3. History of myocardial infarction, stroke, ventricular arrhythmia, or symptomatic conduction abnormality within 12 months.
4. History of congenital QT prolongation.
5. QT >500.
6. Concurrent severe or uncontrolled medical disease (i.e., active systemic infection, diabetes, hypertension, coronary artery disease, congestive heart failure) that, in the opinion of the Investigator, would compromise the safety of the patient or compromise the ability of the patient to complete the study.
7. Symptomatic central nervous system metastases. The patient must be stable after radiotherapy for ≥2 weeks and off corticosteroids for ≥1 week.
8. Pregnant or nursing women.
9. Hypersensitivity or intolerance to Chloroquine, Paclitaxel, Docetaxel, Abraxane, Ixabepilone or other Taxane like drugs.
10. Severe renal insufficiency (CrCl <30mL/min [Cockcroft and Gault]).
11. History of gastrointestinal bleeding, ulceration, or perforation.
12. Concurrent use of potent CYP3A4 inhibitors, such as ketoconazole, itraconazole,clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, and voriconazole.
13. Concurrent use of potent CYP3A4 inducers, such as dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbitol, and St. John's wort.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-09; Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny C Chang, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (3):
- United States (3):
  - Houston Methodist Hospital Cancer Center, Houston, Texas
  - Houston Methodist Hospital Willowbrook, Houston, Texas
  - Houston Methodist Hospital Sugar Land, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: No
to be determined

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 patients were enrolled in the study and 31 patients were evaluated for response.
Groups:
- Chloroquine With Taxane or Taxane-Like (Paclitaxel, Docetaxel, Abraxane, Ixabepilone) Chemotherapy: Chloroquine (250 mg) was given daily orally with either Paclitaxel or Docetaxel or Abraxane or Ixabepilone chemotherapy every 3 weeks (1 cycle) for a maximum of 6 cycles.
  Paclitaxel: Chloroquine 250mg po daily together with Paclitaxel (Taxane) 175 mg/m2 three hours infusion every three weeks.
  Docetaxel: Chloroquine 250mg po daily together with docetaxel 75 mg/m2 administered intravenously over one hour every three weeks
  Abraxane: Chloroquine 250mg po daily together with Abraxane 260 mg/m2 administered intravenously over 30 minutes every three weeks.
  Ixabepilone: Chloroquine 250mg po daily together with Ixabepilone is 40 mg/m2 administered intravenously over three hours every three weeks.
Period: Overall Study
Arm/Group | Chloroquine With Taxane or Taxane-Like (Paclitaxel, Docetaxel, Abraxane, Ixabepilone) Chemotherapy
Started | 38
Completed | 31
Not Completed | 7
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1
Not completed — Toxicity | 3

BASELINE CHARACTERISTICS:
Arm/Group | Chloroquine With Taxane or Taxane-Like (Paclitaxel, Docetaxel, Abraxane, Ixabepilone) Chemotherapy
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 54.1 [31.7 to 78.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38
Metastatic breast cancer [Count of Participants; unit: Participants] | 23
Locally advanced breast cancer [Count of Participants; unit: Participants] | 15
HR+ HEGFR- breast cancer [Count of Participants; unit: Participants] | 20
Triple Negative Breast Cancer [Count of Participants; unit: Participants] | 18

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: To determine the anti-tumor activity of the combination of Chloroquine + Taxane or Taxane-like chemo agents (Paclitaxel, Docetaxel, Abraxane, Ixabepilone) (C/T) measured by overall Response Rate (ORR) defined as percentage of patients having complete or partial response in therapy per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.", or similar definition that is accurate and appropriate.
  The study was designed to compare the ORR with the published percentage of 30% (docetaxel 100 mg/ml2 every 3 weeks for maximum of 10 cycles).
Time Frame: 3-week cycles for maximum of 6 cycles (4.5 months)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chloroquine With Taxane or Taxane-Like (Paclitaxel, Docetaxel, Abraxane, Ixabepilone) Chemotherapy
Number analyzed (Participants) | 31
percentage of participants | 45.16 [29.2 to 62.2]

2. Secondary Outcome: Time to Progression Free Survival (PFS)
Description: To assess the time to progression free survival of patients treated with the combination of Chloroquine and Taxane or Taxane-Like chemotherapy. Progression is defined as time from initiation of chemotherapy to disease progression using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions", or similar definition as accurate and appropriate.
Time Frame: 25.4 months (median)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chloroquine With Taxane or Taxane-Like (Paclitaxel, Docetaxel, Abraxane, Ixabepilone) Chemotherapy
Number analyzed (Participants) | 31
months | 12.4 [4.9 to 24.6]

3. Secondary Outcome: Time of Overall Survival (OS)
Description: To assess the time of overall survival of patients receiving Chloroquine + Taxane or Taxane-like chemotherapy
Time Frame: a median of 25.4 months, up to 83.5 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chloroquine With Taxane or Taxane-Like (Paclitaxel, Docetaxel, Abraxane, Ixabepilone) Chemotherapy
Number analyzed (Participants) | 31
months | 25.4 [13.7 to 83.5]

4. Secondary Outcome: Number of Patients Who Experienced Grade 3 of Greater Adverse Events
Description: To assess how many patients experienced grade 3 or greater adverse events when receiving the combination of Chloroquine and Taxane or Taxane-Like chemotherapy. Toxicity was assessed for all enrolled patients who received one or more doses of the study drug combination by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: 25.4 months (median)
Measure: Count of Participants; unit: Participants
Arm/Group | Chloroquine With Taxane or Taxane-Like (Paclitaxel, Docetaxel, Abraxane, Ixabepilone) Chemotherapy
Number analyzed (Participants) | 31
Participants | 4

ADVERSE EVENTS:
Time Frame: Serious Adverse Events and Other (Not Including Serious) Adverse Events were assessed from time of informed consent up to 30 months. All-Cause Mortality was assessed up to 85 months and reported at a median follow-up of 25.36 months.
Arm/Group | Chloroquine With Taxane or Taxane-Like (Paclitaxel, Docetaxel, Abraxane, Ixabepilone) Chemotherapy
All-Cause Mortality (participants affected / at risk) | 21/31
Serious Adverse Events (participants affected / at risk) | 1/38
Other Adverse Events (participants affected / at risk) | 9/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chloroquine With Taxane or Taxane-Like (Paclitaxel, Docetaxel, Abraxane, Ixabepilone) Chemotherapy (N=38)
Neutropenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chloroquine With Taxane or Taxane-Like (Paclitaxel, Docetaxel, Abraxane, Ixabepilone) Chemotherapy (N=38)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Back pain (General disorders) | 1
Dehydration (General disorders) | 1
Fatigue (General disorders) | 2
Infusion reaction (General disorders) | 1
Syncope (General disorders) | 1
Hand-foot syndrome (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-07-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT01446016/Prot_SAP_000.pdf